CLINICAL TRIAL: NCT00070291
Title: A Phase II Study of Cyclosporine in the Treatment of Angioimmunoblastic T-Cell Lymphoma
Brief Title: Cyclosporine in Treating Patients With Recurrent or Refractory Angioimmunoblastic T-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000331864; U10CA021115 (NIH); E2402 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: angioimmunoblastic T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Immunoblastic Lymphadenopathy | interventions — Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclosporine (Experimental): High dose cyclosporine weeks 1-6, then maintenance dose cyclosporine weeks 7-36. If CR, PR, or SD at week 36 evaluation, treatment is complete. If progression occurs during weeks 7-36, patients will re-register to Step 2 at time of PD and begin high dose therapy (weeks 1-6), followed by maintenance therapy (weeks 7-36). At second progression patients will end protocol treatment.
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: cyclosporine — Cyclosporine doses will be based on actual body weight unless actual body weight is > 15 kg higher than the ideal body weight. Cyclosporine dose will be adjusted to maintain a trough whole blood level of 250-450 ng/mL during the high dose period (weeks 1 -6, starting dose will begin at cyclosporine 3 mg/kg by mouth two times a day (PO BID)) and 150-250 ng/mL during the maintenance period (weeks 7-36, maintenance dose will begin at cyclosporine 2 mg/kg PO BID) in the absence of renal toxicity
  Other Names: CSA,; Neoral,; Gengraf

SUMMARY:
RATIONALE: Cyclosporine may help the immune system slow the growth of angioimmunoblastic T-cell lymphoma.

PURPOSE: This phase II trial is studying how well cyclosporine works in treating patients with recurrent or refractory angioimmunoblastic T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (complete and partial) in patients with recurrent or refractory angioimmunoblastic T-cell lymphoma treated with cyclosporine.

Secondary

* Determine the disease-free, progression-free, and overall survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: Patients receive oral cyclosporine twice daily for up to 36 weeks in the absence of unacceptable toxicity or disease progression during weeks 1-6. Patients experiencing disease progression during weeks 7-36, receive an additional 36 weeks of therapy.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of angioimmunoblastic T-cell lymphoma (recurrent or refractory) based on histologic examination.
* At least one objective measurable or evaluable disease parameter.
* Have failed at least one type of treatment: chemotherapy, auto-transplant, or steroid treatment. Patients may not receive concurrent chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate renal function as indicated by creatinine <= 1.5 the upper limit of normal (ULN).
* Adequate liver function as indicated by alkaline phosphatase, Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) <= 2x the upper limit of normal.
* Total bilirubin <= 2x the upper limit of normal.
* Age 18 or older.

Exclusion Criteria:

* Prior cyclosporine or Tacrolimus (FK506).
* Prior allogeneic transplant.
* Evidence of active infection.
* Congestive heart failure, kidney failure, liver failure, or other severe co-morbidities.
* Evidence of active neurological impairment.
* Previous history of hypersensitivity to cyclosporine and/or Cremorphor EL (polyoxyethylated oil).
* History of other malignancies (other than cured carcinomas in situ of the cervix or basal cell carcinoma of the skin).
* pregnant or breastfeeding women.
* Human immunodeficiency virus (HIV) positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-01-24 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjana Advani, MD, Study Chair — Stanford University
Locations (23):
- United States (23):
  - Stanford Cancer Center, Stanford, California
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Hematology Oncology Associates of Illinois - Berwyn, Berwyn, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - St. Rita's Medical Center, Lima, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between September 2, 2005 and March 24, 2009. The first patient was accrued on January 24, 2006. The study was terminated due to slow accrual.
Groups:
- Cyclosporine: Cyclosporine doses will be based on actual body weight unless actual body weight is > 15 kg higher than the ideal body weight. Cyclosporine dose will be adjusted to maintain a trough whole blood level of 250-450 ng/mL during the high dose period (weeks 1 -6) and 150-250 ng/mL during the maintenance period (weeks 7-36) in the absence of renal toxicity.
  High dose cyclosporine weeks 1-6, then maintenance dose cyclosporine weeks 7-36. If CR, PR, or SD at week 36 evaluation, treatment is complete. If progression occurs during weeks 7-36, patients will re-register to Step 2 at time of PD and begin high dose therapy (weeks 1-6), followed by maintenance therapy (weeks 7-36). At second progression patients will end protocol treatment.
Period: Step 1
Arm/Group | Cyclosporine
Started | 4
Treated | 3
Completed | 2
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Period: Step 2
Arm/Group | Cyclosporine
Started | 1 (One patient completed step 1, but opted to get alternative therapy. One patient entered step 2.)
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cyclosporine
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial Response)
Description: Response was assessed based upon the criteria from the International Workshop to Standardize Criteria for Non-Hodgkin's Lymphoma. Response included complete response and partial response. Complete response was defined as complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related B-symptoms if present prior to therapy, as well as normalization of those biochemical abnormalities definitely attributed to NHL. All lymph nodes and nodal masses must have regressed to normal size. Partial response was defined as a decrease of > 50% in the SPD (sum of the products of the diameters) of the six largest (or less) dominant nodes or nodal masses, no increase in the size of the liver or the spleen, and no new sites of disease.
Time Frame: Assessed at weeks 6, 12, 24 and 36 from onset of treatment, and then at 1 year, 18 months, 2 years and 3 years from registration during follow-up.
Population: all 4 enrolled patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Cyclosporine
Number analyzed (Participants) | 4
Proportion of participants | 0.25 [0.007 to 0.81]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from randomization to death from any cause.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 1 year.
Population: all 4 enrolled patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cyclosporine
Number analyzed (Participants) | 4
Months | 36 [5 to 36]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | Cyclosporine
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=3)
Hematologic-other (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=3)
Anemia (Blood and lymphatic system disorders) | 1
Leukopenia (Leukocytes, decreased) (Investigations) | 2
Neutropenia (Neutrophils, decreased) (Investigations) | 1
Thrombocytopenia (Platelets, decreased) (Investigations) | 1
Hematologic-other (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 1
Edema limb (General disorders) | 2
Creatinine, increased (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Metabolic/Laboratory-other (Investigations) | 2
Neuropathy-sensory (Nervous system disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Head/headache (Nervous system disorders) | 2
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No